CLINICAL TRIAL: NCT04069312
Title: Roflumilast or Azithromycin to Prevent COPD Exacerbations (RELIANCE)
Acronym: RELIANCE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00179281
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe; Chronic Bronchitis
Keywords: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; COPD; Roflumilast; Daliresp; Azithromycin
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast; Azithromycin

STUDY DESIGN:
Intervention Model Description: The trial is a parallel, pragmatic non-inferiority trial with two treatment groups, roflumilast and azithromycin. Up to 1,250 participants will be randomized (1:1) to receive a prescription for one of the two treatments. Treatment assignments will be stratified by site and smoking status (former versus current) using a permuted block design with multiple block sizes.
Masking Description: Treatment assignments will be concealed prior to randomization. Once a patient is assigned to receive a treatment, the clinician, Site Coordinator and patient will not be masked. i.e., they will know the treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast arm (Active Comparator): Participants will receive prescription for Roflumilast (250 mcg/day x 4 weeks, then 500 mcg/day or alternate regimen) x 6 to 72 months
  Interventions: Drug: Roflumilast
- Azithromycin arm (Active Comparator): Participants will receive prescription for Azithromycin (250 mg/day, or 500 mg three times per week, or alternate regimen) x 6 to 72 months
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Roflumilast — Prescription for Roflumilast (250 mcg/day x 4 weeks, then 500 mcg/day or alternate regimen) x 6 to 72 months
  Other Names: Daliresp
  Arms: Roflumilast arm
Drug: Azithromycin — Prescription for Azithromycin (250 mg/day, or 500 mg three times per week, or alternate regimen) x 6 to 72 months
  Other Names: Zithromax
  Arms: Azithromycin arm

SUMMARY:
A multi-center, randomized, 72-month, parallel- group, non-inferiority, phase III study to compare the effectiveness of roflumilast (Daliresp, 500 mcg quaque die (QD) or alternate regimen) therapy versus azithromycin (250 mg QD, 500 mg QD three times per week, or alternate regimen) to prevent hospitalization or death in a patients at high risk for COPD exacerbations.

DETAILED DESCRIPTION:
RELIANCE is a U.S.-based pragmatic clinical trial funded by the Patient-Centered Outcomes Research Institute (PCORI) to compare long-term use of roflumilast vs. azithromycin in up to 1,250 patients. It is intended to support hospital efforts to reduce the risk of all-cause hospitalization and reduce pre-mature deaths in individuals with chronic obstructive pulmonary disease (COPD) who have been hospitalized in the prior year for a COPD exacerbation. The COPD Patient Powered Research Network (PPRN) and affiliated investigators will conduct the trial in sites in the U.S.

Both roflumilast and azithromycin have been shown to reduce the risk of COPD exacerbations compared to placebo. However, there has not been a head-to-head comparison of the two medications. So, the relative harms and benefits of the two medications are unknown. Eligible patients will be randomized (1:1) to receive either a prescription for roflumilast or a prescription for azithromycin, and will be followed for at least 6 and up to 72 months. The primary endpoint is the combined outcome of all-cause hospitalization or death; the secondary endpoints include premature treatment discontinuation, patient-reported adverse effects, and physical, social, and emotional health. Patients will be enrolled at participating clinical sites and follow up data will be collected via an online patient portal or via a call center. Baseline and outcome data will also be collected from site medical records and administrative/claims databases.

Pragmatic, non-inferiority trial using an intention-to-treat analysis to evaluate whether daily azithromycin is non-inferior to daily roflumilast in patients at high risk of COPD exacerbations. The investigators will randomize individual patients to receive prescriptions for roflumilast or azithromycin (1:1 ratio), stratified by site and current smoking status (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* Patient and treating clinician considering treatment intensification with roflumilast or azithromycin to reduce the risk of COPD exacerbations
* Age ≥ 40 years
* Current or past smoker of at least 10 pack-years
* Diagnosis by treating physician of severe COPD and associated chronic bronchitis
* Hospitalized with a diagnosis of COPD exacerbation or respiratory complications due to COVID 19 in the past 12 months
* Current medications include inhaled Long Acting Muscarinic Antagonist (LAMA), Long Acting Beta Agonist (LABA) /LAMA, or Inhaled Corticosteroids (ICS) /LABA(note patients prescribed or using SABA, SAMA, or SABA/SAMA on a scheduled basis (e.g., every 6 hours) are eligible since the patient is receiving functional controller therapy);
* English or Spanish speaking
* Willing and able to provide a contact telephone number.

Exclusion Criteria:

* Unable or declines to provide informed consent;
* Declines to provide social security number, health insurance claims number or Tax Payer ID (as applicable)
* History of intolerance to azithromycin or roflumilast that the patient or patient's treating clinician considers sufficiently serious to avoid either treatment option;
* Current treatment with long-term (more than 30 days) roflumilast, azithromycin or ensifentrine (previous treatment with 1 or more doses of azithromycin, roflumilast or ensifentrine is not an exclusion criterion, as long as the patient and clinician are seeking treatment intensification options and would be willing to use azithromycin or roflumilast, as per randomized treatment assignment.)
* Known hypersensitivity to azithromycin, erythromycin, any macrolide or ketolide antibiotic;
* History of cholestatic jaundice/hepatic dysfunction associated with prior use of azithromycin
* Moderate to severe liver impairment (Child-Pugh B or C)
* Current pregnancy
* Any other clinician-determined exclusion as per the clinician's clinical practice
* The clinicians will be provided the FDA-approved prescribing information for roflumilast and azithromycin. The prescribing information includes a list of warnings and precautions that identifies the potential for adverse effects and is intended to support clinical decision-making that takes into account the risks and benefits of roflumilast and azithromycin for each patient

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of All-cause hospitalizations | Up to 72 months
  All-cause hospitalizations
Number of All-cause deaths | Up to 72 months
  All-cause deaths

SECONDARY OUTCOMES:
Number of All-cause individual events | Up to 72 months
  All-cause individual events
Change in physical function as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) scale | Baseline, 3 months, 6 months and every 6 months up to 72 months
  Based on the scoring scale; a score of 5 is the most favorable and a score of 1 is least favorable.
Change in problems with sleep as assessed by the PROMIS scale | Baseline, 3 months, 6 months and every 6 months up to 72 months
  1 is least favorable and 5 is most favorable
Change in fatigue as assessed by the PROMIS scale | Baseline, 3 months, 6 months and every 6 months up to 72 months
  0 is most favorable and 4 and least favorable
Change in anxiety as assessed by the PROMIS scale | Baseline, 3 months, 6 months and every 6 months up to 72 months
  Score of 1 is most favorable and 5 is least favorable
Change in depression as assessed by the PROMIS scale | Baseline, 3 months, 6 months and every 6 months up to 72 months
  1 is most favorable and 5 is least favorable
Number of Adverse Events | Up to 72 months
  Adverse events
Medication Adherence as assessed by patient self-report | Up to 72 months
  Medication Adherence will be assessed by self-report via Call Center or Patient Portal; Medicare claims data in a subset.
Number of participants that switch to alternate study medication | Up to 72 months
  Patient will be assigned either azithromycin or roflumilast at randomization. We will assess any switch to either roflumilast from azithromycin or azithromycin from roflumilast by self-report via Call Center or Patient Portal, query of clinic staff; Medicare claims data in a subset
Out of pocket cost for study medication | Up to 72 months
  Out of pocket costs for roflumilast of azithromycin by self-report via Call Center or Patient Portal
Change in weight | 3 and 6 months
  Weight in lbs
Number of participants that discontinued medication | Up to 72 months
  This will be collected by self-report via Call Center or Patient Portal; query of clinic staff; Medicare claims data in a subset

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Krishnan, MD, PhD, Principal Investigator — University of Illinois Chicago; Robert Wise, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (29):
- United States (29):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California, Davis Health, Sacramento, California
  - Northwestern, Chicago, Illinois
  - University of Illinois, Chicago, Chicago, Illinois
  - NorthShore Hospital, Glenview, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Baystate Health, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Missouri, Kansas City, Kansas City, Missouri
  - Northern Westchester Hospital/Northwell Health, Mount Kisco, New York
  - Mount Sinai, New York, New York
  - Lenox Hill Hospital/Northwell Health, New York, New York
  - University of North Carolina, School of Medicine, Chapel Hill, North Carolina
  - Duke, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Kaiser Permanente, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Baylor Scott & White (BSW) Health-North, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - Providence Health and Services, Spokane, Washington